CLINICAL TRIAL: NCT01671488
Title: BrUOG 276: A Phase I/II Evaluation of ADXS11-001, Mitomycin,5-fluorouracil (5-FU) and IMRT for Anal Cancer
Brief Title: A Phase I/II Evaluation of ADXS11-001, Mitomycin, 5-fluorouracil (5-FU) and IMRT for Anal Cancer
Acronym: 276
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: pilot data to be used for upcoming larger trial.
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Principal Investigator, howard safran, Principal Investigator, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 276
Record Dates: First submitted 2012-08-07; First posted 2012-08-23 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Anal Cancer
Keywords: Anal Cancer; Mitomycin; 5-Fluorouracil; 5-FU; IMRT; ADXS11-001
MeSH Terms: conditions — Anus Neoplasms | interventions — Therapeutics; Fluorouracil; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): The first dose will be given 10-14 days prior to the initiation of chemoradiation.
  Patient will then receive 5-FU: 1 gm/m2/day x 96 hours beginning on day 1-4 and day 29-32 + 7 days and Mitomycin: 10 mg/m2, day 1 and 29 with IMRT radiation: 54 Gy in 30 fractions at 1.8 Gy per fraction.
  The 2-4th dosages of ADXS11-001 will not be until after completion of all chemoradiation. The second dosage of ADXS11-001 will not be administered until a minimum of 10 days after completion of chemoradiation. The subsequent third and fourth treatment with of ADXS11 will be administered at 28 day intervals.
  Interventions: Biological: Treatment; Drug: 5FU; Drug: Mitomycin; Radiation: IMRT

INTERVENTIONS:
Biological: Treatment — ADXS11-001 will be given at a dose of 1x109 cfu intravenously once every 28 days for 4 total doses. All 4 doses of ADXS11-001 will be 1x109 cfu.
  Other Names: ADXS11-001
Drug: 5FU — 1 gm/m2/day x 96 hours beginning on day 1-4 and day 29-32 + 7 days
Drug: Mitomycin — 10 mg/m2, day 1 and 29 (day 29 can be + 7 days)
Radiation: IMRT — 54 Gy in 30 fractions at 1.8 Gy per fraction.

SUMMARY:
The main purpose of this study is to study the safety and effectiveness of ADXS11-001 when combined with standard chemotherapy and radiation treatment for anal cancer. ADXS11-001 is an investigational agent that is not approved by the FDA to treat anal cancer or any other cancer.

DETAILED DESCRIPTION:
Novel treatments are needed in anal cancer. An important percentage of patients with locally advanced anal cancer will have persistent loco-regional disease or develop systemic metastases. Virtually all cases of anal cancer are related to infection by HPV. Anal cancer cells infected with HPV have the tumor associated antigen HPV E7. ADXS11-001 causes antigen presenting cells to be stimulated to facilitate immune cells to attack cancer cells expressing HPV E7. ADXS11-001, at the phase II dose of 1x109 CFU, has been shown to be safe in patients with advanced cervical cancer which also is caused by HPV infection. Anti-tumor activity and safety have been demonstrated in cervical cancer to single agent ADXS11-001 and the combination of ADXS11-001 and cisplatin chemotherapy. Data presented at ASCO 2012 ADXS11-001 is currently being evaluated in women in the United States with cervical intraepithelial neoplasia. Radiation may augment the activity of ADXS11-001 increasing the exposure of tumor related antigens thereby increasing the chance for loco-regional disease eradication and preventing systemic recurrence. Therefore, ADXS11-001 may increase complete response, prevent recurrence disease and increase disease-free and overall survival in anal cancer. This protocol will develop sufficient preliminary safety and efficacy data to facilitate the investigation of ADXS11-001 in anal cancer within "NRG", the newly formed cooperative group based on the merger of the RTOG, NSABP and GOG.

As described above, Phase I studies and preliminary data from phase II studies have demonstrated that ADXS11-001, 1x109 CFU, can be safely administered as a single agent and in combination with chemotherapy. For example in over 200 patients treated at the dose of 1x109CFU there have been no cases of severe listeria bacteremia or grade 3 cardiopulmonary toxicity. However, since ADXS11-001 has not previously been administered with radiation, the primary objective of this study will be to establish the safety of the addition of ADXS11-001 to chemoradiation for anal cancer. The following schedules will be assessed.

• Treatment Schedule: The first dose will be given 10-14 days prior to the initiation of chemoradiation. The 2nd-4th dosages of ADXS11-001will not be until after completion of all chemoradiation. The second dosage of ADXS11-001 will not be administered until a minimum of 10 days after completion of chemoradiation, ANC > 1,000 cells/mm3, serum creatinine < 1.5 mg/dl and all toxicities from chemoradiation have resolved to grade 2 or less. The subsequent third and fourth treatment with of ADXS11 will be administered at 28 day intervals. This will provide the needed safety data to evaluate Treatment Schedule #2.

Standard treatment with mitomycin, 5-FU and radiation for anal cancer has substantial toxicity. In RTOG 9811, 74% of patients had grade 3/4 nonhematologic toxicity and 61% of patients had grade 3 or grade 4 hematologic toxicity from this regimen. Therefore, the toxicities of standard chemoradiation with mitomycin, 5-FU and radiation are well above the conventionally accepted parameters in a phase I study even prior to adding ADXS11-001. However, it is critical that the addition of ADXS-11-001 does not compromise the delivery of potentially curative standard chemoradiation for anal cancer.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Histologically-proven, invasive primary squamous, basaloid, or cloacogenic carcinoma of the anal canal; 3.1.2 AJCC 2009 TN Stage: T1N1-N3, T2(< 4cm)N1-N3, T2(> 4cm)N0,T3N0-3, T4N0-3;based upon the following minimum diagnostic workup: 3.1.2.1 History/physical examination within 14 days prior to registration; 3.1.2.2 Within 42 days prior to registration, the patient must have an anal examination by any of the following: colonoscopy, sigmoidoscopy, or rigid proctoscopy, with documentation of primary anal lesion size, distance from anal verge.

3.1.3 Groin examination within 42 days prior to registration with documentation of any groin adenopathy and lymphadenopathy (location: right vs. left; medial vs. lateral; mobile vs. fixed; and size); 3.1.4 X-ray (PA and lateral), CT scan, or PET/CT scan of the chest within 42 days prior to registration; 3.1.5 CT scan, MRI, or PET/CT of the abdomen and pelvis within 42 days prior to registration; 3.1.6 Zubrod Performance Status 0-1; 3.1.7 Age ≥ 18; 3.1.8 Laboratory data obtained ≤ 14 days prior to registration on study, with adequate bone marrow, hepatic and renal function defined as follows:

* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3;
* Platelets ≥ 100,000 cells/mm3;
* Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.);
* Serum creatinine ≤ 1.5 mg/dl;
* Bilirubin < 1.4mg/dl;
* ALT/AST < 3 x ULN;
* Negative serum pregnancy test for women of child-bearing potential; 3.1.9 Women of childbearing potential and male participants must agree to use a 2 forms of medically effective means of birth control (such as a condom and spermicide) throughout their participation in the treatment phase of the study and for 90 days post last dose of study drug.

3.1.10 Patients must sign a study-specific informed consent prior to study entry.

3.1.11 Patients with a history of clinically significant pulmonary disease must have PFTs demonstrating a DLCO ≥ 40%. This testing is considered standard of care prior to mitomycin, 5-FU and radiation.

3.1.12 Patients with a history of clinically significant cardiac disease must have a LVEF ≥ 30% by ECHO. (MUGA scan may also be used to determine LVEF) This testing is considered standard of care prior to mitomycin, 5-FU and radiation.

3.1.13 Patients must be able to swallow pills.

Exclusion Criteria:

3.2.1 Prior invasive malignancy (except non-melanomatous skin cancer), unless disease free for a minimum of 2 years; 3.2.2 Prior systemic chemotherapy for anal cancer; 3.2.3 Prior allergic reaction to the study drugs involved in this protocol. 3.2.4 Prior radiotherapy to the pelvis that would result in overlap of radiation therapy fields; 3.2.5 Severe, active co-morbidity, defined as follows: 3.2.5.1 Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris and cardiac arrhythmia are ineligible. Furthermore, patients with unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months are ineligible; 3.2.5.2 Patients with active infection requiring systemic therapy (oral or IV) or those currently receiving antibiotics that cannot discontinue prior to dosing are ineligible.

3.2.5.3 Transmural myocardial infarction within the last 6 months; 3.2.5.4 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; 3.2.5.5 Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration; 3.2.5.6 Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; 3.2.6 Patients known to be seropositive for HIV and/or active hepatitis, even if liver function studies are in the eligible range.

3.2.7 Other immunocompromised status (e.g., organ transplant or chronic glucocorticoid use).If patient has diagnosis of immunodeficiency, is dependent on or has received systemic steroids therapy or any form of immunosuppressive therapy within 7 days prior to the first dose of ADXS11-001 they are ineligible. Topical corticosteroid or occasional inhaled corticosteroids are allowed.

3.2.8 Women who are pregnant or lactating are ineligible because the treatment involved in this study may be significantly teratogenic and there is the potential for transmission of listeria to the infant.

3.2.9 Patients allergic to or with a sensitivity to penicillin, ampicillin, trimethoprim-sulfa and quinolones (including history of rash or anaphylaxis).

3.2.10 Patients allergic to naproxen. 3.2.11 Patients receiving oral or IV antibiotics 3.2.12 Patients with a prior history of a splenectomy and/or sickle cell trait/disease 3.2.13 Patient has implanted medical device(s) that pose a high risk for colonization and/or cannot be easily removed (e.g., prosthetic joints, artificial heart valves, pacemakers, orthopedic screw(s), metal plate(s), bone graft(s), or other exogenous implant(s)). NOTE: More common devices and prosthetics which include arterial and venous stents, dental and breast implants and venous access devices (e.g. Port-a-Cath or Mediport) are permitted. Sponsor must be contacted prior to consenting any subject who has any other device and/or implant. Site is required to submit to BrUOG ALL surgical implants patient has ever had in their medical history and ALL surgeries regardless of link to this cancer diagnosis.

3.2.14 Patients who are receiving or may receive future treatment with PI3K or TNFα inhibitors. To be confirmed by treating medical oncologist in writing 3.2.15 Has undergone a major surgery, including surgery for a new artificial implant and/or device, within 6 weeks prior to the initiation of ADXS11-001 treatment. NOTE: if patient underwent surgery > 6 weeks from start of ADSX11-001, all toxicities and/or complications must have recovered to baseline or Grade 1 prior to the initiation of ADXS11-001 study therapy.

3.2.16 Patient not being willing to have new infusion line placed for each infusion of ADXS11-001 as existing or newly placed central venous catheter or infusion ports are not allowed to be used for ADXS11-001 administration. Must be confirmed as discussed with patient and that they agreed.

3.2.17 Patient not willing to comply with requirement of central venous catheter or infusion port must not be used for 72 hours following the completion of the ADXS11-001 infusion and the patient receives the first post-treatment dose of oral antibiotics. Must be confirmed as discussed with patient and that they agreed.

3.2.18 Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed. All recent vaccines (within 30 days) to be listed on conmed log 3.2.19 Patient has a history of listeriosis or prior ADXS11-001 therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Brown University
Locations (3):
- United States (3):
  - Montefiore Medical Center, New York, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: The first dose will be given 10-14 days prior to the initiation of chemoradiation.
  Patient will then receive 5-FU: 1 gm/m2/day x 96 hours beginning on day 1-4 and day 29-32 + 7 days and Mitomycin: 10 mg/m2, day 1 and 29 with IMRT radiation: 54 Gy in 30 fractions at 1.8 Gy per fraction.
  The 2-4th dosages of ADXS11-001 will not be until after completion of all chemoradiation. The second dosage of ADXS11-001 will not be administered until a minimum of 10 days after completion of chemoradiation. The subsequent third and fourth treatment with of ADXS11 will be administered at 28 day intervals.
  Treatment: ADXS11-001 will be given at a dose of 1x109 cfu intravenously once every 28 days for 4 total doses. All 4 doses of ADXS11-001 will be 1x109 cfu.
  5FU: 1 gm/m2/day x 96 hours beginning on day 1-4 and day 29-32 + 7 days
  Mitomycin: 10 mg/m2, day 1 and 29 (day 29 can be + 7 days)
  IMRT: 54 Gy in 30 fractions at 1.8 Gy per fraction.
Period: Overall Study
Arm/Group | Treatment
Started (This is for patients who signed consent) | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 60.36 [37 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Safety of the Addition of ADXS11-001 to Standard Chemoradiation for Patients With Anal Cancer.
Description: Evaluate maximal toxicities via CTCAE version 4.0 All adverse events, serious and non-serious, were captured from date of ICF through 4 weeks post treatment completion- regardless of causality.
Time Frame: Baseline, then prior to each ADXS11-001 and weekly during radiation. Assessments 1-2 weeks post radiation then 2-6 weeks post vaccine and off study and 30 days post treatment.
Population: Patient's who received treatment on study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: To Evaluate the 6-month Clinical Complete Response Rate for Patients With Anal Cancer Treated With ADXS11-001 Mitomycin, 5-FU and IMRT.
Description: Patients to undergo tumor evaluation assessment (via sigmoidoscopy, proctoscopy, colonoscopy or anoscope) 6 months post the start of chemotherapy/radiation.
Time Frame: Tumor evaluation 6 months after coming off study
Population: Number of patient's who received treatment on study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 10
Participants | 9

3. Secondary Outcome: To Evaluate Progression-free and Overall Survival for Patients With Anal Cancer Treated With ADXS11-001, Mitomycin, 5-FU and IMRT.
Description: Patients terminating study treatment early prior to disease recurrence will be followed every 6 months for year 1 then annually for a total of 5 years. The follow-up portion will commence once patient comes off study or post the 2-6 week post the 4th treatment time point/visit.
  Assessments were tumor evaluation via sigmoidoscopy, proctoscopy, colonoscopy or anoscope and also chest/abdomen/pelvic imaging.
Time Frame: Follow up and survival status at 6 months and 1 year post coming off study and annually until patient has been off for 5 years
Population: As one patient expired prior to 6 month assessment, the total n used was 9 to assess PFS
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 9
Participants | 8

ADVERSE EVENTS:
Time Frame: SAEs and AEs are captured from the time of consent until 30 days post the last treatment. SAEs occurring post 30 days are required to be reported if they are potentially related.
Description: Please note that all SAEs and AEs that occurred and were reported are noted in this database, but that does not mean that the SAEs or AEs reported here in the results table are related to the study drug ADXS11-001 or the combination. In short, these are SAEs or AEs that occurred, but the reporting of them here, does not equate to a relationship to study treatment.
  The SAEs include multiple events but this represents the actual SAE as reported by the site and as reported to NIH OBA and the FDA.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 10/10
Serious Adverse Events (participants affected / at risk) | 10/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=10)
fever (1), hypotension(2) (Investigations) | 1 (1)
fever (1), hypotension(2) Hypokalemia (3) (Investigations) | 1 (1)
weakness (3), decreased appetite (2), GI bleed(3). Anemia(3) (Investigations) | 1 (1)
Nausea (3), dehydration (3), anal mucositis (3), enterocolitis (2) (Investigations) | 1 (1)
Nausea(3),dehydration(3),anal mucositis(3), (Investigations) | 1 (1) — enterocolitis(2),colitis(2),perianal pain(3), diarrhea(2),weakness(2),Anemia(2)
Expired unknown reason (5) (Investigations) | 1 (1)
seizure (3), catastrophic pulmonary or cardiac event or massive CVA (5) (Investigations) | 1 (1)
PLT(4), diarrhea (2), ANC (3), fever (1) (Investigations) | 1 (1)
Diarrhea (3), dehydration(3), wt loss (2), back pain (2), fatigue (2), (Investigations) | 1 (1) — hypokalemia (3), HGB(3), PLT (2), Glucose (1), Hyponatremia (1), albumin(1), hypocalcemia (1), WBC (2), Lymph (4)
Diarrhea (2), wt loss (2) , back pain (1), fatigue (2), (Investigations) | 1 (1) — HGB(2), PLT (3), Glucose-hyperglycemia (1), , albumin(2), hypocalcemia (2), WBC (2), Lymph (2), fever (2)
fever (1) headache (1) (Investigations) | 1 (1)
Fever(1*)febrile neutropenia(3*)ANC(3*)WBC (4*), PLT (4*) (Investigations) | 1 (1) — Anemia (3*)cellulitis (2*)acute kidney injury(2*)creatinine(2*)mucositis(1*)Lymph(4*)
ANC (4*)WBC(4*)PLT(3*)Anemia (3*)cellulitis (2*),mucositis (1*)Lymph (4*), (Investigations) | 1 (1) — thromboembolic event(2*),left lower leg edema(1*)
chest pain (1*), shortness of breath (3*), lightheadedness (1*) (Investigations) | 1 (1)
Rectal bleeding (3*), Anemia (2*) , ANC(3*) , PLT(4*) , Fever (1*) (Investigations) | 1 (1) — Dermatitis radiation (3*) , pain rectal (2*)
Rectal bleeding (3*)Anemia (3*)ANC(4*)PLT(4*)Fever (1*) (Investigations) | 1 (1) — Dermatitis radiation (3*)pain rectal (2*)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=10)
allergies (Investigations) | 2 (2)
ALT (Investigations) | 2 (2)
anal mucositis (Investigations) | 1 (1)
ANC (Investigations) | 2 (2)
Anemia (Investigations) | 3 (3)
anorexia (Investigations) | 2 (2)
anxiety (Investigations) | 1 (1)
APTT (Investigations) | 1 (1)
AST (Investigations) | 2 (2)
chills/rigors (Investigations) | 8 (8)
constipation (Investigations) | 2 (2)
confusion (Investigations) | 1 (1)
creatinine (Investigations) | 1 (1)
Dehydration (Investigations) | 2 (2)
depression (Investigations) | 2 (2)
Diarrhea (Investigations) | 5 (5)
Frequent stools (non-diarrhea) (Investigations) | 1 (1)
fecal incontinence (Investigations) | 2 (2)
Dizziness (Investigations) | 3 (3)
dyspepsia (Investigations) | 1 (1)
Dyspnea/SOB (Investigations) | 3 (3)
edema (Investigations) | 2 (2)
erythoderma/erythema (Investigations) | 1 (1)
dry skin (Investigations) | 1 (1)
ejaculatory dysfunction (Investigations) | 1 (1)
epistaxis (Investigations) | 1 (1)
Fatigue (Investigations) | 6 (6)
fever (Investigations) | 3 (3)
flu-like symptoms (Investigations) | 1 (1)
gastritis (Investigations) | 1 (1)
GI bleed/bloody diarrhea/rectal bleed (Investigations) | 1 (1)
H/A (Investigations) | 5 (5)
hematuria (Investigations) | 2 (2)
Hot flashes (Investigations) | 3 (3)
Hyperpigmentation (Investigations) | 2 (2)
hyperglycemia (Investigations) | 1 (1)
Hypoalbumin (Investigations) | 4 (4)
Hypocalcemia (Investigations) | 2 (2)
hypohydrosis (Investigations) | 1 (1)
HypoK (Investigations) | 5 (5)
HypoMG (Investigations) | 2 (2)
Hyponatremia (Investigations) | 8 (8)
hypotension (Investigations) | 1 (1)
Hypertension (Investigations) | 5 (5)
INR (Investigations) | 1 (1)
Lightheadedness (Investigations) | 1 (1)
lymphocyte decrease (Investigations) | 7 (7)
migraine (Investigations) | 1 (1)
mucositis/mouth sores (Investigations) | 8 (8)
myalgia (Investigations) | 2 (2)
arthralgia (Investigations) | 2 (2)
nausea (Investigations) | 7 (7)
pain-abdomen (Investigations) | 4 (4)
pain/back and neck (Investigations) | 3 (3)
pain secondary to abcess/infection (Investigations) | 1 (1)
pain-epigastric (Investigations) | 1 (1)
pain-general (Investigations) | 1 (1)
pain-joints (Investigations) | 1 (1)
pain-leg (Investigations) | 2 (2)
rectal pain/perianal pain (Investigations) | 5 (5)
paresthesia (Investigations) | 2 (2)
PLT (Investigations) | 5 (5)
Radiation Dermatitis (Investigations) | 4 (4)
rash (Investigations) | 1 (1)
skin ulceration/Groin sore (Investigations) | 3 (3)
infection (cellulitis/small intestine, abscess, UTI, vaginal) (Investigations) | 3 (3)
social circumstances (Investigations) | 1 (1)
sore throat (Investigations) | 1 (1)
Tachycardia (Investigations) | 1 (1)
tooth infection (Investigations) | 1 (1)
urinary frequency (Investigations) | 1 (1)
urinary pain/dysuria (Investigations) | 3 (3)
urinary retention (Investigations) | 1 (1)
vomitng (Investigations) | 3 (3)
WBC (Investigations) | 6 (6)
weakness (Investigations) | 1 (1)
wt loss (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT01671488/Prot_SAP_ICF_000.pdf